CLINICAL TRIAL: NCT04334707
Title: Kidney Precision Medicine Project
Acronym: KPMP
Status: Recruiting | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Michigan (Other); Icahn School of Medicine at Mount Sinai (Other); Brigham and Women's Hospital (Other); Broad Institute of MIT and Harvard (Other); The Cleveland Clinic (Other); Columbia University (Other); European Molecular Biology Laboratory (Unknown); Indiana University (Other); Johns Hopkins University (Other); Joslin Diabetes Center (Other); Pacific Northwest National Laboratory (U.S. Federal Agency); Princeton University (Other); Stanford University (Other); Ohio State University (Other); University of California, San Diego (Other); University of California, San Francisco (Other); University of Pittsburgh (Other); The University of Texas Health Science Center at San Antonio (Other); University of Texas (Other); Washington University School of Medicine (Other); Yale University (Other)
Responsible Party: Principal Investigator, Jonathan Himmelfarb, Professor, School of Medicine, University of Washington
Other Study IDs: SITE00000750; U2CDK114886 (NIH); UH3DK114861 (NIH); UH3DK114866 (NIH); UH3DK114870 (NIH); UH3DK114908 (NIH); UH3DK114915 (NIH); UH3DK114926 (NIH); UH3DK114907 (NIH); UH3DK114920 (NIH); UH3DK114923 (NIH); UH3DK114933 (NIH); UH3DK114937 (NIH)
Record Dates: First submitted 2020-03-23; First posted 2020-04-06 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Acute Kidney Failure; Acute Kidney Insufficiency; Acute Renal Failure; Acute Renal Injury; Acute Renal Insufficiency; Kidney Failure, Acute; Kidney Insufficiency, Acute; Renal Failure, Acute; Renal Insufficiency, Acute; Chronic Kidney Diseases; Chronic Kidney Insufficiency; Chronic Renal Diseases; Chronic Renal Insufficiency; Kidney Insufficiency, Chronic
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency, Chronic | interventions — Laparotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Kidney (renal) tissue will be obtained from all study participants at study entry Blood and urine will be collected longitudinally, including DNA One-time stool sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute Kidney Injury Cohort: The focus will be on acute intrinsic non-glomerular disease, primarily on acute tubular necrosis (ATN). KPMP will also include a special population of patients at risk for AKI or with early AKI captured by an open (surgical) kidney biopsy performed at the time of clinically indicated laparotomy.
  Interventions: Procedure: Kidney Biopsy
- Chronic Kidney Diseases Cohort: High priority populations include CKD in the setting of diabetes (diabetic kidney disease, DKD) and hypertension-associated CKD (H-CKD). A special population of people with long-standing type 1 diabetes (more than 25 years) who remain free of clinically-evident DKD will also be included.
  Interventions: Procedure: Kidney Biopsy

INTERVENTIONS:
Procedure: Kidney Biopsy — A kidney biopsy is a procedure that involves taking a small piece of kidney tissue for examination with a microscope. A licensed health care provider will perform a kidney biopsy.
  Other Names: Renal Biopsy; Laparotomy

SUMMARY:
Acute kidney injury (AKI) and chronic kidney disease (CKD) impose a significant global health burden. Yet, no effective therapies currently exist for AKI, and only a few are available for CKD.

Despite significant effort from industry and academia, development of pharmacologic therapies for AKI and CKD has been hampered by:

Non-predictive animal models The inability to identify and prioritize human targets The limited availability of human kidney biopsy tissue A poor understanding of AKI and CKD heterogeneity Historically, AKI and CKD have been described as single, uniform diseases. However, growing consensus suggests that different disease pathways lead to different subgroups of AKI and CKD (AKIs and CKDs).

Access to human kidney biopsy tissue is a critical first step to define disease heterogeneity and determine the precise molecular pathways that will facilitate identification of specific drug targets and ultimately enable individualized care for people with AKI and CKD.

A number of research centers across the United States are collaborating to bring state-of-the-art technologies together to:

* Ethically obtain and evaluate kidney biopsies from participants with AKI or CKD
* Define disease subgroups
* Create a kidney tissue atlas
* Identify critical cells, pathways, and targets for novel therapies

The KPMP is made up of three distinct, but highly interactive, activity groups:

* Recruitment Sites: The recruitment sites (RS) are responsible for recruiting participants with AKI or CKD into the longitudinal study and performing the kidney biopsy.
* Tissue Interrogation Sites: The tissue interrogation sites (TIS) are responsible for developing and using innovative technologies to analyze the biopsy tissue.
* Central Hub: The central hub is responsible for aggregating, analyzing, and visualizing the generated data and providing scientific, infrastructure, and administrative support for the KPMP consortium.

DETAILED DESCRIPTION:
The Kidney Precision Medicine Project (KPMP) is a prospective cohort study, whose goal is to use deep molecular phenotypes of kidney biopsies, along with longitudinally collected clinical phenotypic data, in order to develop new disease ontologies, classification systems, and treatments for acute kidney injury (AKI) and chronic kidney disease (CKD). Since its inception, the KPMP has sought out and included substantive patient-representative feedback regarding disease experience, lack of innovation in new kidney disease therapies and patient tolerance for risk levels in balance with potential benefits both to the individual and society.

The KPMP Has publicly and operationally committed itself to always put participants and their best interests first and this foundational principle informs and undergirds every facet of the study. Both AKI and CKD are conditions that impose a significant global health burden. Yet, no effective therapies currently exist for AKI, and only a few are available for CKD. The network will utilize state-of-the-art methods to perform molecular interrogation of the tissue and to link the molecular data to kidney structure and clinical information in the form of a kidney tissue atlas.

Molecular and imaging data derived from kidney tissue will be integrated with clinico-pathologic and genetic information, as well as other data derived from analyses of fluid biospecimens, including peripheral blood, urine, and stool. Using advanced analytics to integrate the data, KPMP will aim to define kidney disease subgroups in molecular terms by identifying critical cells, pathways and targets for novel therapies.

Patients with AKI or CKD will be recruited from clinical care encounters (e.g., clinic visits for CKD patients, hospitalization or emergency room visits for AKI patients) and from electronic resources (e.g., existing registries, electronic health records). All study procedures are designed to optimize participant safety and will be ethically conducted, ensuring subjects fully understand the scope of the study and any possible risks.

For each participant, kidney tissue will be obtained for molecular phenotyping and clinical diagnosis. The diagnostic interpretation will be returned to the participant's primary caregiver to inform clinical care, but no treatment interventions will be prescribed by the KPMP. In addition to kidney biopsy, the study will involve collection of baseline (time of biopsy) and longitudinal biospecimens (including urine, plasma, serum, DNA and stool) and demographic, clinical, and laboratory data. Participants will be followed through scheduled in-person and remote (telephone) study visits, as well as through periodic review of electronic health records.

ELIGIBILITY:
Chronic Kidney Disease Subjects Inclusion Criteria Diabetic kidney disease (DKD)

* Diagnosis of diabetes mellitus (type 1 or 2) established by at least one of the following criteria:

  * Hemoglobin A1C greater than or equal to 6.5%, confirmed with a repeat test within the past year
  * Fasting blood sugar greater than or equal to 126 mg/dL, confirmed with a repeat test within the past year
  * Use of glucose-lowering therapy (insulin or oral or other subcutaneous agents)
  * International Classification of Diseases (ICD) 9/10 diagnostic code for diabetes
* Evidence of persistent kidney damage, manifest as any of the following present on at least two clinic assessments prior to enrollment and at least 3 months apart and excluding subjects with acute medical illnesses and changing kidney function:

  * Estimated glomerular filtration rate 30-59 mL/min/1.73m2
  * Estimated glomerular filtration rate greater than or equal to 60 mL/min/1.73m2 with urine albumin excretion greater than or equal to 30 mg/g creatinine (or mg/day)
  * Estimated glomerular filtration rate greater than or equal to 60 mL/min/1.73m2 with urine protein excretion greater than or equal to 150 mg/g creatinine (or mg/day)

Hypertension-associated Chronic Kidney Disease (H-CKD) Inclusion Criteria

* Diagnosis of hypertension (HTN) established by at least one of the following criteria:

  * BP greater than 140/90 mmHg measured on three occasions over at least 1 month
  * Taking antihypertensive medication for blood pressure (BP) control
  * International Classification of Diseases (ICD) 9/10 diagnostic code for hypertension
* Evidence of persistent kidney damage, manifested as any of the following present on at least two assessments at least 3 months apart and excluding subjects with acute medical illnesses and changing kidney function:

  * Estimated glomerular filtration rate 30-59 mL/min/1.73m2 on two assessments at least 3 months apart with albuminuria or proteinuria less than 2000 mg/g creatinine (or mg/day)
  * Estimated glomerular filtration rate greater than or equal to 60 mL/min/1.73m2 with urine albumin excretion 30-2000 mg/g creatinine (or mg/day)
  * Estimated glomerular filtration rate greater than or equal to 60 mL/min/1.73m2 with urine protein excretion 150-2000 mg/g creatinine (or mg/day)

Acute Kidney Injury Subjects Inclusion Criteria

All three of the following criteria must be met:

* Baseline estimated glomerular filtration rate greater than 45 mL/min/1.73m2. Baseline defined by the median of the last three outpatient serum creatinine measurements from day 7 to 365 prior to enrollment.

  * If only two measurements obtained within this window, the two results will be averaged.
  * If only one measurement was obtained within this window, this result will be used
  * If baseline is missing the potential participant can be enrolled with an estimated baseline, but only if there is no past medical history of chronic kidney disease.
* Elevated serum creatinine (greater than or equal to 1.5 times baseline as defined above).
* And at least ONE of the following:

  * A repeat serum creatinine within 48 hours of initial serum creatinine, showing a further increase of 0.3 mg/dL
  * Positive kidney injury urine biomarker, as defined by any of the following:

    * NGAL level greater than or equal to 150 ng/mL by ELISA or clinical analyzer
    * KIM1 level greater than or equal to 2.8 ng/mL by ELISA
    * TIMP2 x IGFBP7 greater than or equal to 2.0 by NephroCheck®
  * Urine microscopy suggestive of acute tubular necrosis defined as a urine microscopy score of greater than or equal to 2.

    * greater than or equal to 1 Renal Tubular Epithelial cells (RTE) per high powered field (HPF) AND greater than or equal to 1 granular cast/ low powered field (LPF); or
    * greater than or equal to 5 Renal Tubular Epithelial cells (RTE) per high powered field (HPF); or
    * greater than or equal to 5 granular cast/ low powered field (LPF)

General Exclusion Criteria:

* Under 18 years of age
* Body Mass Index (BMI) greater than 40 kg/m2
* Allergy to iodinated contrast (any reaction)
* Pregnancy
* Malignancy - Receiving active chemotherapy or radiation to treat malignancy (except for nephrectomy tissue for reference and feasibility studies)
* Transplant recipient (includes solid transplant and bone marrow)
* Additional vulnerable individuals (incarcerated, institutionalized, or otherwise unable to participate in the study)
* Inability to provide informed consent
* Clinical diagnosis of kidney disease from an autoimmune disease, dysproteinemia, viral disease or glomerular disease other than DKD or H-CKD
* Unwilling to receive blood transfusion (if needed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The KPMP will focus on participant populations that account for large proportions of the public health burden of acute and chronic kidney diseases as evidenced by research and federal data.
  For CKD, high priority populations include CKD in the setting of diabetes (diabetic kidney disease, DKD) and hypertension-associated CKD (H-CKD). A special population of people with long-standing type 1 diabetes (more than 25 years) who remain free of clinically-evident DKD will also be included.
  For AKI, the focus will be on acute intrinsic non-glomerular disease, primarily on acute tubular necrosis (ATN). KPMP will also include a special population of patients at risk for AKI or with early AKI captured by an open (surgical) kidney biopsy performed at the time of clinically indicated laparotomy. The rationale for including this special AKI population is that AKI often occurs early in the clinical course of conditions like sepsis, major surgery and trauma.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Biopsy-related outcomes | Immediately after the procedure for up to 6 months
  Biopsy-related complications will be collected by KPMP study staff using standardized case report forms. Clinical utility of the biopsy results will be assessed using standardized surveys of clinical providers, and participant-reported outcomes will be assessed using standardized questionnaires. Biopsy-related outcomes data will be collected around the time of the biopsy and within the six months following procurement of the kidney biopsy.
Kidney disease progression outcomes | Through study completion (up to 10 years, depending on enrollment date of participant)
  Longitudinal change in estimated glomerular filtration rate (eGFR):
  * Primary composite longitudinal outcome, defined by any of the following:
  * ESRD, defined as initiation of maintenance dialysis or kidney transplantation
  * Sustained decline in eGFR by 40% or more from baseline
  * Individual components of the primary composite outcome
  * Slope of eGFR change (from baseline to the latest value)
Kidney disease progression outcomes | Through study completion (up to 10 years, depending on enrollment date of participant)
  Longitudinal change in urine albumin excretion defined by the following:
  -Slope of change in urine albumin-creatinine ratio
Kidney disease progression outcomes | Through study completion (up to 10 years, depending on enrollment date of participant)
  Longitudinal change in urine albumin excretion defined by the following:
  -Change of Kidney Disease Improving Global Outcomes (KDIGO) albuminuria stage

OTHER OUTCOMES:
Number of Participants with Additional Outcome Measures | Through study completion (up to 10 years, depending on enrollment date of participant)
  * All-cause mortality, defined by death from any cause and validated through linkages with the National Death Index (NDI)
  * Cardiovascular events, including heart failure, myocardial infarction, cerebrovascular event, transient ischemic attack, thromboembolic event, arrhythmia, and cardiac arrest
  * New AKI events after KPMP enrollment
  * Hospital admissions and discharge diagnoses after KPMP enrollment
Number of Participants with Outcomes Specific to AKI | Through study completion (up to 10 years, depending on enrollment date of participant)
  * Duration of AKI: number of days with elevated serum creatinine above baseline
  * Recovery of AKI: return of serum creatinine to greater than 125% of baseline by 3 months post-biopsy
  * ICU admissions: admissions to any intensive care unit during hospitalization
  * Need for dialysis: initiation and duration of any dialysis modality (CRRT, HD, or PD)
  * Length of hospital stay: number of days during initial AKE episode

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Himmelfarb, MD, Principal Investigator — University of Washington
Locations (8):
- United States (8):
  - Yale University, New Haven, Connecticut
  - Johns Hopkins University, Baltimore, Maryland
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Joslin Diabetes Center, Boston, Massachusetts
  - Columbia University, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas at Southwestern, Dallas, Texas

REFERENCES:
- [Background] USGAO, Kidney disease research funding and priority setting. 2017: [online] https://www.gao.gov/assets/690/681714.pdf.
- [Background] RM, B., Social security amendments of 1972: summary and legislative history. 1973
- [Background] Rettig RA. Special treatment--the story of Medicare's ESRD entitlement. N Engl J Med. 2011 Feb 17;364(7):596-8. doi: 10.1056/NEJMp1014193. No abstract available. PMID 21323539
- [Background] Norris KC, Williams SF, Rhee CM, Nicholas SB, Kovesdy CP, Kalantar-Zadeh K, Ebony Boulware L. Hemodialysis Disparities in African Americans: The Deeply Integrated Concept of Race in the Social Fabric of Our Society. Semin Dial. 2017 May;30(3):213-223. doi: 10.1111/sdi.12589. Epub 2017 Mar 9. PMID 28281281
- [Background] Prevention, C.f.D.C.a., National Chronic Kidney Disease Fact Sheet, 2017, U.D.o.H.a.H. Services, Editor. 2017: Atlanta, GA.
- [Background] Mendu ML, Erickson KF, Hostetter TH, Winkelmayer WC, Olan G, Meyer RN, Hakim R, Sedor JR. Federal Funding for Kidney Disease Research: A Missed Opportunity. Am J Public Health. 2016 Mar;106(3):406-7. doi: 10.2105/AJPH.2015.303009. No abstract available. PMID 26885959
- [Background] Linde PG, Archdeacon P, Breyer MD, Ibrahim T, Inrig JK, Kewalramani R, Lee CC, Neuland CY, Roy-Chaudhury P, Sloand JA, Meyer R, Smith KA, Snook J, West M, Falk RJ. Overcoming Barriers in Kidney Health-Forging a Platform for Innovation. J Am Soc Nephrol. 2016 Jul;27(7):1902-10. doi: 10.1681/ASN.2015090976. Epub 2016 Apr 28. PMID 27127187
- [Background] Inrig JK, Califf RM, Tasneem A, Vegunta RK, Molina C, Stanifer JW, Chiswell K, Patel UD. The landscape of clinical trials in nephrology: a systematic review of Clinicaltrials.gov. Am J Kidney Dis. 2014 May;63(5):771-80. doi: 10.1053/j.ajkd.2013.10.043. Epub 2013 Dec 6. PMID 24315119
- [Background] Hsu RK, McCulloch CE, Dudley RA, Lo LJ, Hsu CY. Temporal changes in incidence of dialysis-requiring AKI. J Am Soc Nephrol. 2013 Jan;24(1):37-42. doi: 10.1681/ASN.2012080800. Epub 2012 Dec 6. PMID 23222124
- [Background] Lameire NH, Bagga A, Cruz D, De Maeseneer J, Endre Z, Kellum JA, Liu KD, Mehta RL, Pannu N, Van Biesen W, Vanholder R. Acute kidney injury: an increasing global concern. Lancet. 2013 Jul 13;382(9887):170-9. doi: 10.1016/S0140-6736(13)60647-9. Epub 2013 May 31. PMID 23727171
- [Background] Collister D, Pannu N, Ye F, James M, Hemmelgarn B, Chui B, Manns B, Klarenbach S; Alberta Kidney Disease Network. Health Care Costs Associated with AKI. Clin J Am Soc Nephrol. 2017 Nov 7;12(11):1733-1743. doi: 10.2215/CJN.00950117. Epub 2017 Oct 19. PMID 29051143
- [Background] Kellum JA, Bellomo R, Ronco C. Kidney attack. JAMA. 2012 Jun 6;307(21):2265-6. doi: 10.1001/jama.2012.4315. No abstract available. PMID 22572776
- [Background] USRDS, United States Renal Data Systems 2013 Annual Data Report. United States Renal Data Systems. 2013: [online] http://http://www.usrds.org/2013/pdf/v1_ch6_13.pdf.
- [Background] Waikar SS, Liu KD, Chertow GM. Diagnosis, epidemiology and outcomes of acute kidney injury. Clin J Am Soc Nephrol. 2008 May;3(3):844-61. doi: 10.2215/CJN.05191107. Epub 2008 Mar 12. PMID 18337550
- [Background] Sileanu FE, Murugan R, Lucko N, Clermont G, Kane-Gill SL, Handler SM, Kellum JA. AKI in low-risk versus high-risk patients in intensive care. Clin J Am Soc Nephrol. 2015 Feb 6;10(2):187-96. doi: 10.2215/CJN.03200314. Epub 2014 Nov 25. PMID 25424992
- [Background] Murugan R, Karajala-Subramanyam V, Lee M, Yende S, Kong L, Carter M, Angus DC, Kellum JA; Genetic and Inflammatory Markers of Sepsis (GenIMS) Investigators. Acute kidney injury in non-severe pneumonia is associated with an increased immune response and lower survival. Kidney Int. 2010 Mar;77(6):527-35. doi: 10.1038/ki.2009.502. Epub 2009 Dec 23. PMID 20032961
- [Background] Coca SG, Yusuf B, Shlipak MG, Garg AX, Parikh CR. Long-term risk of mortality and other adverse outcomes after acute kidney injury: a systematic review and meta-analysis. Am J Kidney Dis. 2009 Jun;53(6):961-73. doi: 10.1053/j.ajkd.2008.11.034. Epub 2009 Apr 5. PMID 19346042
- [Background] Waikar SS, Winkelmayer WC. Chronic on acute renal failure: long-term implications of severe acute kidney injury. JAMA. 2009 Sep 16;302(11):1227-9. doi: 10.1001/jama.2009.1364. No abstract available. PMID 19755705
- [Background] Coca SG, Singanamala S, Parikh CR. Chronic kidney disease after acute kidney injury: a systematic review and meta-analysis. Kidney Int. 2012 Mar;81(5):442-8. doi: 10.1038/ki.2011.379. Epub 2011 Nov 23. PMID 22113526
- [Background] Kellum JA, Sileanu FE, Murugan R, Lucko N, Shaw AD, Clermont G. Classifying AKI by Urine Output versus Serum Creatinine Level. J Am Soc Nephrol. 2015 Sep;26(9):2231-8. doi: 10.1681/ASN.2014070724. Epub 2015 Jan 7. PMID 25568178
- [Background] AKIWG, K., Kidney Disease: Improving Global Outcomes (KDIGO) Clinical Practice Guideline for Acute Kidney Injury. Kidney inter., Suppl., 2012. 2: p. 1-138.
- [Background] Chu R, Li C, Wang S, Zou W, Liu G, Yang L. Assessment of KDIGO definitions in patients with histopathologic evidence of acute renal disease. Clin J Am Soc Nephrol. 2014 Jul;9(7):1175-82. doi: 10.2215/CJN.06150613. Epub 2014 May 1. PMID 24789552
- [Background] Perazella MA, Coca SG, Hall IE, Iyanam U, Koraishy M, Parikh CR. Urine microscopy is associated with severity and worsening of acute kidney injury in hospitalized patients. Clin J Am Soc Nephrol. 2010 Mar;5(3):402-8. doi: 10.2215/CJN.06960909. Epub 2010 Jan 14. PMID 20089493
- [Background] Corapi KM, Chen JL, Balk EM, Gordon CE. Bleeding complications of native kidney biopsy: a systematic review and meta-analysis. Am J Kidney Dis. 2012 Jul;60(1):62-73. doi: 10.1053/j.ajkd.2012.02.330. Epub 2012 Apr 24. PMID 22537423
- [Background] Rodriguez LL, Brooks LD, Greenberg JH, Green ED. Research ethics. The complexities of genomic identifiability. Science. 2013 Jan 18;339(6117):275-6. doi: 10.1126/science.1234593. No abstract available. PMID 23329035
- [Result] CfMaM., S., Chronic Conditions among medicare beneficiaries. Chartbook, 2012 Edition. Baltimore 2012.